CLINICAL TRIAL: NCT03817645
Title: Pilot-trial on the Use of the Panaceo Medicine Product "MED" for the Treatment of IBS (Irritable Bowel Syndrome)
Brief Title: Panaceo "MED" for IBS (Irritable Bowel Syndrome)
Acronym: PCeo-17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scigenia GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCeo-17
Record Dates: First submitted 2018-12-19; First posted 2019-01-25 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Irritable Bowel Syndrome; Microbial Colonization; Intestinal Disease
Keywords: Zeolite
MeSH Terms: conditions — Irritable Bowel Syndrome; Communicable Diseases; Intestinal Diseases | interventions — Zeolites

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Panaceo MED (Experimental): Zeolite, Medicinal product, class IIa for oral intake, daily intake of 2 sachets (3 g), for 3 months.
  Interventions: Other: Zeolite
- Control (Placebo Comparator): Micro crystalline cellulose daily intake of 2 sachets (3 g), for 3 months.
  Interventions: Other: Zeolite

INTERVENTIONS:
Other: Zeolite — The natural zeolite clinoptilolite is of volcanic origin. The mineral belongs to the group of zeolite minerals. Zeolites are silicates with a microporous structure. This results in a stable structure with nanometer-sized cavities that pass through the natural zeolite clinoptilolite - comparable to a mineral sponge. Due to the numerous pores and channels, the mineral has a large internal surface and it can absorb molecules that are smaller in diameter than the pore openings. Since zeolite clinoptilolite has an anionic charge, there are cations such as Na +, K +, Ca 2+, Mg 2+ which can be exchanged for other ions (e.g., Pb^2+) in the cavities for electrical charge balance. In particular, the ion exchange capacity is essential for the effect and is used in many areas.

SUMMARY:
Zeolite clinoptilolite is a volcanic mineral from the group of zeolites. The porous structure is associated with a large inner surface. Due to the anionic framework charge, ions (e.g., Pb^2+) can be absorbed or exchanged. The specific Panaceo PMA zeolite is approved as a class IIa medical device for the repair of the intestine inner lining. It is CE certified and complies with the relevant European Union regulations in terms of safety and effectiveness. Zeolite is known for its absorbing properties. Because of these properties and the results of several human studies, it warrants the investigation of possible effects on specific indications in human medicine, e.g. irritable bowel syndrome.

The diagnosis "irritable bowel syndrome (IBS)" is according to the ROME Foundation, an US medical society. IBS is a disorder with dysfunction of the bowels, a latent inflammation is discussed. The present study aims to evaluate the following effects in patients with IBS:

* Primary endpoint: effect on the symptoms of IBS.
* Secondary endpoint: intestinal wall permeability, integrity of the tight junctions as measured by the change in zonulin concentration in the stool.
* Further endpoints:

  * Inflammation parameters and anti-inflammatory laboratory parameters.
  * Biodiversity of the gastrointestinal microbiome.
  * histamine-associated parameters.
  * Constipation as a possible side effect.

For this purpose, a double-blind randomized controlled trial (RCT) is realized prospectively in a monocentric outpatient-controlled study. The subjects take the test compound daily (verum, reference substance) for 12 weeks and document the intake of the study-substance, intake of medications, stool-frequency and consistency. They receive "before" and "after" the intervention phase a blood and stool analysis for the determination of parameters for intestinal wall integrity (zonulin) inflammation (hsCRP, interleukin-10, calprotectin), histamine metabolism, microbiome diversity. The pilot study is realized ahead of the detailed planning of a later main study.

ELIGIBILITY:
Inclusion Criteria:

* Frequency of discomfort or pain in the abdomen in the last 3 months, more than 1 day per week.
* Start of the discomfort or pain more than 6 months ago.
* Improvement of the discomfort or pain associated with bowel movements sometimes, often, frequently, always.
* Association of the discomfort or pain with a frequency change in bowel movements sometimes, often, frequently, always.
* Association of the discomfort or pain with a change in stool-consistency sometimes, often, frequently, always.

Exclusion Criteria:

* Age: younger than 18, older than 80.
* Diagnosed inflammatory bowel disease (M. Crohn, Colitis Ulcerosa)
* Diagnosed nutritional idiosyncrasy
* Cancer treatment in the last 12 weeks
* Depression in the last 12 weeks
* Intake of weight loss supporting medication (Lipase inhibitors)
* Alcohol, nicotine, drug-abuse
* Status after organ-transplantation, intake of immunosuppressants
* Acute or chronic neurologic or psychiatric disease
* Acute or chronic heart disease or kidney disease
* Acute or chronic liver damage or any other organ damages
* Transient severe obstipation in the last 4 weeks
* Transient acute diarrhea in the last 4 weeks (e.g. intestinal infection)
* Intestinal cancer
* Intake of Panaceo MED or other Zeolite in the last 4 weeks
* Type I Diabetes or severe metabolic disease
* Infection with fever in the last 4 weeks
* Intake of cortisone or antibiotics in the last 4 weeks
* Planed journey of more than 14 days in the next 12 weeks (change of nutritional habits)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Abdominal discomfort or pain | 3 months
  Frequency: 0 - never, 1 - less than once / month, 2 - once / month, 3 - two-three days / month, 4 - once per week, 5 - more than once per week, 6 - every day.
Symptom improvement with defaecation | 3 months
  0 - never or rarely, 1 - sometimes, 2 - often, 3 - frequently, 4 - always.
Stool frequency associated with abdominal discomfort or pain (more or less frequent) | 3 months
  0 - never or rarely, 1 - sometimes, 2 - often, 3 - frequently, 4 - always.
Stool consistency associated with abdominal discomfort or pain (softer or harder) | 3 months
  0 - never or rarely, 1 - sometimes, 2 - often, 3 - frequently, 4 - always.

SECONDARY OUTCOMES:
Stool laboratory parameter: Firmicutes | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Prevalence Firmicutes (CFU/g stool)
Stool laboratory parameter: Bacteroidetes | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Prevalence Bacteroidetes (CFU/g stool)
Stool laboratory parameter: Ratio: Bacteroidetes/Firmicutes | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Computation of Ratio: Bacteroidetes/Firmicutes
Stool laboratory parameter: Butyrat Producers | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Prevalence of Butyratproducing bacteria (CFU/g stool)
Stool laboratory parameter: Clostridia | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Prevalence of Clostridia (CFU/g stool)
Stool laboratory parameter: Histaminproducers, | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Prevalence of Histaminproducing bacteria (CFU/g stool)
Stool laboratory parameter: H2S producers | 3 months
  Genotyping of bacteria in stool, before and after intake of study substance; Prevalence of H2S-producing bacteria (CFU/g stool)

OTHER OUTCOMES:
Change of permeability (Leaky-Gut) | 3 months
  Zonulin (< 55 ng/ml) in stool
Change of bowel inflammation | 3 months
  Calprotectin (< 50 mg/l) in stool
Change of permeability of mucosa | 3 months
  Alpha 1-Antitrypsin (< 27,5 mg/dl) in stool
Change of the inflammation mediator | 3 months
  Histamin (< 600 ng/ml) in stool
Efficacy of binding and elimination of ammoniak | 3 months
  Ammoniak (11-51 µmol/l) in blood / serum
Change of inflammation | 3 months
  high sensitivity C-reactive protein (mg/l) in blood / serum
Change of anti-inflammatory mediator | 3 months
  Interleukin-10 (< 9,1 pg/ml) in blood / serum
Possible release of metal ions | 3 months
  Aluminium (< 11 µg/l) in blood / serum
Change of histamin metabolism | 3 months
  Di-Amino-Oxydase (> 10 U/ml) in blood / serum

CONTACTS AND LOCATIONS:
Overall Officials: Ventzislav Petkov, M.D., Principal Investigator — Physician
Locations (1):
- SCIgenia GmbH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamprecht M, Bogner S, Steinbauer K, Schuetz B, Greilberger JF, Leber B, Wagner B, Zinser E, Petek T, Wallner-Liebmann S, Oberwinkler T, Bachl N, Schippinger G. Effects of zeolite supplementation on parameters of intestinal barrier integrity, inflammation, redoxbiology and performance in aerobically trained subjects. J Int Soc Sports Nutr. 2015 Oct 20;12:40. doi: 10.1186/s12970-015-0101-z. eCollection 2015. PMID 26500463